CLINICAL TRIAL: NCT04701476
Title: An Open Label Phase II Study for the Treatment of Liver Metastatic Colorectal Cancer and Non-Small Cell Lung Cancer With a Combination of TATE (Trans-Arterial Tirapazamine Embolization) and Pembrolizumab
Brief Title: TATE and Pembrolizumab (MK3475) in mCRC and NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teclison Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT-007; KEYNOTE-A91 (Other: Merck & Co.)
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Lung Cancer
Keywords: colorectal cancer; NSCLC; pembrolizumab; tirapazamine; Liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms | interventions — pembrolizumab; trifluridine tipiracil drug combination; regorafenib

STUDY DESIGN:
Intervention Model Description: Open-label study in two indications. The mCRC cohort will be a randomized trial for TATE+Pembrolizumab versus standard 3rd line therapy for mCRC. The NSCLC cohort will be single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- colorectal cancer (Experimental): metastatic colorectal cancer progressed on at least two lines of chemotherapy
  Interventions: Drug: TATE and pembrolizumab; Drug: TAS-102 pill; Drug: Regorafenib Pill
- NSCLC (Experimental): Liver metastatic NSCLC progressed on immune checkpoint inhibitors and chemotherapy
  Interventions: Drug: TATE and pembrolizumab

INTERVENTIONS:
Drug: TATE and pembrolizumab — All liver metastatic lesions will be treated with TATE for maximally debulking. Pembrolizumab IV infusion per standard schedule every 3 or 6 weeks until progression or maximally 2 years.
  Other Names: TATE: Trans-arterial Tirapazamine Embolization;
Drug: TAS-102 pill — The comparator of the mCRC arm is TAS-102 at 60 mg BID 5 days per week for 2 weeks then 2 weeks off.
  Other Names: LONSURF
  Arms: colorectal cancer
Drug: Regorafenib Pill — As an alternative to TAS-102 per treating physician's discretion. If selected, Regorafenib 160 mg oral daily for 3 weeks on and one week off, every 4 weeks per cycle. Do not take Regoarefnib if taking TAS-102.
  Other Names: STIVARGA
  Arms: colorectal cancer

SUMMARY:
Patients with refractory metastatic colorectal cancer or non-small cell lung cancer with liver metastasis treated with Trans-arterial Tirapazamine Embolization along with Pembrolizumab.

DETAILED DESCRIPTION:
This study is an open-label study to treat patients with refractory metastatic colorectal cancer and non-small cell lung cancer with liver metastasis. Patients enrolled in the mCRC cohort will be randomized to receive study treatment Trans-arterial Tirapazamine Embolization (TATE)+Pembrolizumab or FDA-approved standard of care, such as TAS-102 or regorafenib, and their Overall Survival (OS) will be compared in the two cohorts as the primary endpoint. Patients enrolled in the NSCLC cohort will all receive study treatment TATE+Pembrolizaumb and Overall Response Rate (ORR) will be the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Liver metastatic MSS-mCRC or NSCLC without EGFR or AKT mutations
* mCRC progressed on at least two lines of standard chemotherapy; or
* NSCLC progressed on chemotherapy and an immune checkpoint inhibitor
* Measurable disease
* ECOG 0-1
* At least 4 weeks from prior chemotherapy and free from chemo-related toxicity
* Adequate organ function

Exclusion Criteria:

* Prior organ transplantation
* Liver metastasis more than 50%
* Oxygen saturation less than 92% in room air
* Prior autoimmune disorder
* CNS metastasis
* Major GI bleeding in the last 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival for the mCRC cohort | 24 months
  From the first day of treatment to death
Overall Response Rate (ORR) for the NSCLC cohort | within 24 months
  Per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Duration of Response | 24 months
  per RECIST 1.1
Response rate | 24 months
  in TATE treated or TATE-untreated lesions by RECIST and mRECIST
PFS | 24 months
  Progression Free Survival
TTP | 24 months
  Time to Progression

CONTACTS AND LOCATIONS:
Overall Officials: Ray Lee, Study Director — Teclison Limited
Locations (3):
- University of California, Irvine Medical Center, Orange, California, United States
- Taiwan (2):
  - China Medical University Hsinchu Hospital, Hsinchu
  - Chung Shan Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No
International meeting report or medical Journal publication